CLINICAL TRIAL: NCT03333863
Title: Bacterial and Antimicrobial Susceptibility Profile and the Prevalence of Different Sites of Infection in Shengjing Hospital of China Medical University: a Retrospective, Descriptive Study
Brief Title: Bacterial and Antimicrobial Susceptibility Profile and the Prevalence of Different Sites of Infection(BASPP)
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Hongyu Zhao, Clinical Professor, Shengjing Hospital
Other Study IDs: BASPP
Record Dates: First submitted 2017-10-28; First posted 2017-11-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Infectious Diseases in Pneumonia,Nephropyelitis,Angiocholitis or Others; Positive Bacterial Cultures Results of the Medical Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive study which reviewed the data of patients hospitalized with positive bacterial cultures — A retrospective, descriptive study was conducted at shengjing hospital of China Medical University between 2015- 2017. Data regarding bacterial culture isolates, antimicrobial susceptibility spectrum, and the general data of patients with fever or suspicion of sepsis were collected.

SUMMARY:
Positive results of bacterial culture are analyzed comprehensively in Shengjing Hospital of China Medical University in recent 3 years（between 2015- 2017）

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pneumonia, nephropyelitis, angiocholitis or other infectious diseases
* Positive results of bacterial cultures in blood, urine, sputum, and secretion
* The medical records of shengjing hospital of China Medical University from January 2015 to December 2017

Exclusion Criteria:

* Negative results of bacterial cultures in blood, urine, sputum, and secretion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized with positive bacterial cultures results in blood, urine, sputum, and secretion, are enrolled at shengjing hospital of China Medical University from January 2015 to December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1889 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
bacterial and antimicrobial susceptibility profile | From January 2015 to December 2017
  Primary outcome was recording the results of bacterial and antimicrobial susceptibility profile of pneumonia, nephropyelitis, or angiocholitis, measured with statistical methods.

SECONDARY OUTCOMES:
patient's critical condition | From January 2015 to December 2017
  Secondary outcome was evaluating the patient's critical condition, measured with APACHE (acute physiology and chronic health evaluation) II score.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhao, doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musicha P, Cornick JE, Bar-Zeev N, French N, Masesa C, Denis B, Kennedy N, Mallewa J, Gordon MA, Msefula CL, Heyderman RS, Everett DB, Feasey NA. Trends in antimicrobial resistance in bloodstream infection isolates at a large urban hospital in Malawi (1998-2016): a surveillance study. Lancet Infect Dis. 2017 Oct;17(10):1042-1052. doi: 10.1016/S1473-3099(17)30394-8. Epub 2017 Aug 14. PMID 28818544